CLINICAL TRIAL: NCT03873493
Title: A Prospective, Open-Label, Single-Arm, Phase 2, Multicenter Study Evaluating the Efficacy of Venetoclax Plus Ibrutinib in Subjects With T-Cell Prolymphocytic Leukemia
Brief Title: A Study Evaluating the Efficacy of Venetoclax Plus Ibrutinib in Participants With T-cell Prolymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-803; 2018-002179-17 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Leukemia; T-cell Prolymphocytic Leukemia (T-PLL); Cancer
Keywords: T-cell Prolymphocytic Leukemia (T-PLL); Cancer; Venetoclax; Venclexta; Venclyxto; Ibrutinib; Imbruvica; Relapsed or Refractory T-lymphoid malignancy
MeSH Terms: conditions — Leukemia; Leukemia, Prolymphocytic, T-Cell; Neoplasms; Recurrence | interventions — venetoclax; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Ibrutinib (Experimental): Participants received 400 mg venetoclax orally once a day after a 5-day ramp-up and 420 mg ibrutinib orally once a day for up to 2 years or until progressive disease, intolerability, or they became eligible for stem cell transplantation after achieving complete remission.
  Interventions: Drug: Venetoclax; Drug: Ibrutinib

INTERVENTIONS:
Drug: Venetoclax — Venetoclax tablets taken orally once a day (QD). Initially, venetoclax was administered utilizing a 5-step dose ramp-up over 5 days. Subjects were hospitalized and closely monitored for 7 days. The venetoclax ramp-up was administered in a daily manner: 20 mg on Week 1 Day 1, 50 mg on Week 1 Day 2, 100 mg on Week 1 Day 3, 200 mg on Week 1 Day 4, and 400 mg on Week 1 Day 5 and thereafter, once daily, until the end-of-treatment. The dose of venetoclax may have been increased to 600 mg QD at Week 8 or thereafter.
  Other Names: ABT-199; GDC-0199; Venclexta®; Venclyxto®
Drug: Ibrutinib — Ibrutinib capsules taken orally once a day, 420 mg/day until the end-of-treatment.
  Other Names: Imbruvica®

SUMMARY:
The main objective of this study is to evaluate the efficacy of the combination of venetoclax plus ibrutinib for treating adults with T-cell prolymphocytic leukemia (T-PLL).

DETAILED DESCRIPTION:
This study is planned as an adaptive 2-stage design as follows:

Stage 1: Enroll 14 participants with relapsed or refractory (R/R) T-PLL and move to Stage 2 if 4 or more participants meet protocol-specified response criteria. Response assessment will be performed on a continued basis until all 14 participants have enrolled into Stage 1 and have completed the Week 24 disease assessment.

Stage 2: Enroll up to an additional 23 participants.

The study was stopped after Stage 1. Stage 2 was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adequate liver, kidney and hematology function per laboratory values as described in the protocol.
* Diagnosis of T-cell prolymphocytic leukemia (T-PLL) that requires treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Received prior alemtuzumab (unless unsuitable or unavailable).
* Has no malignancies other than T-PLL that:

  * currently require systemic therapies;
  * were not previously treated with curative intention (unless the malignant disease is in a stable remission due to the discretion of the treating physician); or
  * developed signs of progression after curative treatment.

Exclusion Criteria:

* History of or current decompensated cirrhosis including Child-Pugh class B or C, ascites, hepatic encephalopathy, or variceal bleeding.
* Has human T-cell lymphotropic virus, type 1.
* Prior allogeneic stem cell transplant within 6 months of study drug administration and requirement for graft versus host therapy.
* Has an uncontrolled or active infection including severe acute respiratory syndrome- coronavirus-2 (SARS-COV-2).
* Previously treated with a B-cell lymphoma (BCL)-2 inhibitor.
* Received a prohibited therapy within the specified time frame as described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (3):
  - Dana-Farber Cancer Institute /ID# 207728, Boston, Massachusetts
  - Mayo Clinic - Rochester /ID# 207692, Rochester, Minnesota
  - University of Texas MD Anderson Cancer Center /ID# 207746, Houston, Texas
- Peter MacCallum Cancer Ctr /ID# 209554, Melbourne, Victoria, Australia
- Medizinische Universitaet Wien /ID# 208497, Vienna, Vienna, Austria
- Helsinki University Hospital /ID# 208108, Helsinki, Uusimaa, Finland
- France (3):
  - HCL - Hôpital Lyon Sud /ID# 208731, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHRU Lille - Hopital Claude Huriez /ID# 208726, Lille, Hauts-de-France
  - Hopital Pitie Salpetriere /ID# 208730, Paris
- University Hospital Cologne /ID# 208834, Cologne, Germany
- Azienda Sanitaria Universitaria Giuliano Isontina /ID# 211487, Trieste, Italy
- Netherlands (2):
  - Maxima Medisch Centrum /ID# 207989, Eindhoven
  - Universitair Medisch Centrum Groningen /ID# 207990, Groningen
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust /ID# 211264, Oxford, Oxfordshire
  - The Royal Marsden NHS Foundation Trust /ID# 211263, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 16 adults with relapsed or refractory T-cell prolymphocytic leukemia (R/R T-PLL) were screened, and 14 participants were enrolled across 10 sites in 7 countries (Australia, France, Germany, Italy, Netherlands, United Kingdom, and United States).
Pre-assignment Details: This study was planned as an adaptive 2-stage design with Stage 1 to enroll 14 participants and Stage 2 to enroll up to an additional 23 participants based on the number of responders in Stage 1. Results from Stage 1 met the protocol-defined stopping rules, hence Stage 2 was not opened for enrollment. Stage 1 was completed as planned.
  For one participant "study terminated by sponsor" was entered as study discontinuation reason by mistake.
Period: Overall Study
Arm/Group | Venetoclax + Ibrutinib
Started | 14
Completed | 0
Not Completed | 14
Not completed — Withdrawal by Subject | 1
Not completed — Death | 9
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated by Sponsor | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.74)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 0
  40 - < 65 years | 5
  ≥ 65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Disease Duration [Mean (Standard Deviation); unit: years] | 3.229 (3.2134)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was assessed as follows:
  * 0: Fully active, able to carry on all predisease performance without restriction.
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  * 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  * 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  * 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Participants
    0 (Fully active) | 7
    1 (Restricted activity but ambulatory and able to work) | 6
    2 (Ambulatory but unable to work) | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving complete remission (CR), CR with incomplete bone marrow recovery (CRi), or partial remission (PR) as their best response per investigator assessment based on the T-PLL consensus criteria 2019.
  CR: All of the following response criteria must be met:
  Group A:
  * all lymph nodes < 1 cm;
  * spleen < 13 cm;
  * no constitutional symptoms;
  * circulating lymphocyte count < 4 × 10^9/L;
  * bone marrow T-PLL cells < 5% of mononuclear cells;
  * no other specific site involvement
  Group B:
  * platelets ≥ 100 × 10^9 /L;
  * hemoglobin ≥ 11.0 g/dL;
  * neutrophils ≥ 1.5 × 10^9 /L.
  CRi: All of the CR response criteria in Group A met; at least 1 parameter in Group B not achieved, unrelated to T-PLL, but related to drug toxicity.
  PR: At least 2 of the parameters in Group A and 1 parameter in Group B need to improve if previously abnormal. If only 1 parameter of both Groups A and B is abnormal prior to therapy, only 1 parameter needs to improve.
Time Frame: Clinical response was assessed at Weeks 4, 8, 12, 16, and 24 for ORR assessment
Population: The full analysis set includes all participants who received at least 1 dose of study drug (either venetoclax or ibrutinib).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
percentage of participants | 7.1 [0.2 to 33.9]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of first dose of any study drug to the date of earliest disease progression or death. PFS was calculated using Kaplan-Meier methods.
  Response was assessed by the investigator based on the T-PLL consensus criteria 2019.
  Progressive disease (PD) is defined as meeting at least one of the criteria of Group A or Group B below:
  Group A:
  * lymph nodes increase in > 20% in sum of long-axis diameters of up to 3 target lesions (SLD) from nadir;
  * spleen increase ≥ 50% in vertical length beyond normal from baseline;
  * circulating lymphocyte count increase ≥ 50% from baseline;
  * appearance of a new lesion;
  Group B:
  * platelet count decrease of ≥ 50% from baseline due to T-PLL (not due to drug toxicity);
  * hemoglobin decrease of ≥ 2 g/dL from baseline due to T-PLL;
  * neutrophils decrease of ≥ 50% from baseline due to T-PLL.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
months | 2.7 [1.2 to 5.3]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined for participants who achieved a best overall response of CR, CRi, or PR as the time from the date of first response (CR, CRi, or PR) to the earliest date of disease progression or death. DOR was calculated using Kaplan-Meier methods.
  Response was assessed by the investigator based on the T-PLL consensus criteria 2019.
  Progressive disease is defined as meeting at least one of the criteria of Group A or Group B below:
  Group A:
  * lymph nodes increase in > 20% in SLD from nadir;
  * spleen increase ≥ 50% in vertical length beyond normal from baseline;
  * circulating lymphocyte count increase ≥ 50% from baseline;
  * appearance of a new lesion;
  Group B:
  * platelet count decrease of ≥ 50% from baseline due to T-PLL (not due to drug toxicity);
  * hemoglobin decrease of ≥ 2 g/dL from baseline due to T-PLL;
  * neutrophils decrease of ≥ 50% from baseline due to T-PLL.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Full analysis set participants with a best overall response of CR, CRi, or PR
Measure: Median (Full Range); unit: months
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 1
months | 4.6 [4.6 to 4.6]

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from the date of the participant's first dose of any study drug to the date of earliest disease progression. TTP was calculated using Kaplan-Meier methods.
  Clinical response (laboratory and physical examination assessments) was assessed by the investigator according to the T-PLL consensus criteria 2019.
  Progressive disease is defined as meeting at least one of the criteria of Group A or Group B below:
  Group A:
  * lymph nodes increase in > 20% in SLD from nadir;
  * spleen increase ≥ 50% in vertical length beyond normal from baseline;
  * circulating lymphocyte count increase ≥ 50% from baseline;
  * appearance of a new lesion;
  Group B:
  * platelet count decrease of ≥ 50% from baseline due to T-PLL (not due to drug toxicity);
  * hemoglobin decrease of ≥ 2 g/dL from baseline due to T-PLL;
  * neutrophils decrease of ≥ 50% from baseline due to T-PLL.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
months | 2.7 [1.2 to 5.3]

5. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival is defined as time from participant's first dose of any study drug to the date of earliest disease progression, death, or start of a new anti-T-PLL therapy. EFS was calculated using Kaplan-Meier methods.
  Clinical response (laboratory and physical examination assessments) was assessed by the investigator according to the T-PLL consensus criteria 2019.
  Progressive disease is defined as meeting at least one of the criteria of Group A or Group B below:
  Group A:
  * lymph nodes increase in > 20% in SLD from nadir;
  * spleen increase ≥ 50% in vertical length beyond normal from baseline;
  * circulating lymphocyte count increase ≥ 50% from baseline;
  * appearance of a new lesion;
  Group B:
  * platelet count decrease of ≥ 50% from baseline due to T-PLL (not due to drug toxicity);
  * hemoglobin decrease of ≥ 2 g/dL from baseline due to T-PLL;
  * neutrophils decrease of ≥ 50% from baseline due to T-PLL.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
months | 2.6 [0.6 to 5.3]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who achieved CR, CRi, PR, or stable disease (SD) as best overall response per investigator assessment based on the T-PLL consensus criteria 2019.
  Stable disease is defined as meeting all of the following criteria for at least 3 months:
  * lymph nodes change of -29% to +20% in SLD;
  * spleen change of -49% to +49% beyond normal from baseline;
  * circulating lymphocyte count > 30 × 10^9 /L or change of -49% to +49%;
  * platelet count change of -49% to +49%;
  * hemoglobin < 11.0 g/dL or change < 50% from baseline or change < 2 g/dL;
  * neutrophils change of -49% to +49%.
Time Frame: Clinical response was assessed at Weeks 4, 8, 12, 16, and 24 for DCR assessment
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
percentage of participants | 28.6 [8.4 to 58.1]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of the participant's first dose of any study drug to death from any cause. OS was calculated using Kaplan-Meier methods.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
months | 7.3 [1.6 to 10.9]

8. Secondary Outcome: Number of Eligible Participants Reaching Autologous or Allogeneic Transplantation
Description: Participants eligible for autologous or allogeneic transplantation were transplant-naïve participants who achieved CR.
Time Frame: From first dose of study drug to end of study; median time on study was 30.1 weeks.
Population: Participants who were transplant-naive and achieved CR. No participants achieved a CR to be eligible for transplant.
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are any event with onset after the first dose of study drug and no more than 30 days after the last dose of study drug.
  A serious AE was an event that resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, persistent or significant disability/incapacity, or an important medical event requiring medical or surgical intervention to prevent a serious outcome.
  The Investigator rated the severity of each AE according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening and grade 5 = death.
  The Investigator assessed the relationship of the AE to the use of study drug.
Time Frame: From first dose of study drug up to 30 days after last dose; median time on treatment was 13.86 weeks (range 1.0 to 44.4 weeks)
Population: All participants who received at least 1 dose of study drug (either venetoclax or ibrutinib)
Measure: Count of Participants; unit: Participants
Arm/Group | Venetoclax + Ibrutinib
Number analyzed (Participants) | 14
Participants
  Any adverse event | 14
  AE with NCI-CTCAE toxicity Grade 3, 4, or 5 | 11
  Serious adverse event | 8
  AE leading to venetoclax discontinuation, incl PD | 11
  AE leading to venetoclax interruption | 9
  AE leading to venetoclax reduction | 2
  AE with reasonable possibility related to venetoclax | 10
  AE leading to ibrutinib discontinuation, incl PD | 11
  AE leading to ibrutinib interruption | 10
  AE leading to ibrutinib reduction | 1
  AE with reasonable possibility related to ibrutinib | 13
  Serious AE with reasonable possibility related to venetoclax | 3
  Serious AE with reasonable possibility related to ibrutinib | 4
  AE leading to death | 5
  All deaths | 10

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment through the end of study; median time on study was 30.1 weeks. Adverse events are reported from first dose of study drug up to 30 days after last dose; median time on treatment was 13.86 weeks (range 1.0 to 44.4 weeks).
Arm/Group | Venetoclax + Ibrutinib
All-Cause Mortality (participants affected / at risk) | 10/14
Serious Adverse Events (participants affected / at risk) | 8/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Ibrutinib (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 4 (5)
EUTHANASIA (General disorders) | 1 (1)
ASPERGILLUS INFECTION (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 1 (1)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Ibrutinib (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 3 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1)
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 1 (1)
ANDROGEN DEFICIENCY (Endocrine disorders) | 1 (1)
EYE SWELLING (Eye disorders) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 8 (11)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (3)
GLOSSODYNIA (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 6 (7)
PANCREATIC STEATOSIS (Gastrointestinal disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (2)
TONGUE ERUPTION (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)
ASTHENIA (General disorders) | 1 (1)
CATHETER SITE PAIN (General disorders) | 1 (1)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 5 (5)
FATIGUE (General disorders) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
HYPERPLASTIC CHOLECYSTOPATHY (Hepatobiliary disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FOLLICULITIS (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2)
PARVOVIRUS B19 INFECTION (Infections and infestations) | 1 (1)
RHINITIS (Infections and infestations) | 1 (1)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 1 (2)
WOUND (Injury, poisoning and procedural complications) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 (1)
MAGNETIC RESONANCE IMAGING HEAD ABNORMAL (Investigations) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2)
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL ATROPHY (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
DEVICE FAILURE (Product Issues) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2)
BLADDER DIVERTICULUM (Renal and urinary disorders) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (2)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03873493/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03873493/SAP_001.pdf